CLINICAL TRIAL: NCT00683696
Title: Echocardiography Guided Cardiac Resynchronization Therapy (EchoCRT)
Acronym: EchoCRT
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EchoCRT
Record Dates: First submitted 2007-08-30; First posted 2008-05-23 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure; Ventricular Dyssynchrony
Keywords: Cardiac Resynchronization Therapy; Heart Failure; Ventricular Dyssynchrony; Mechanical Dyssynchrony; Intraventricular Dyssynchrony; Echocardiography; Normal QRS; Heart Disease; EchoCRT
MeSH Terms: conditions — Heart Failure; Heart Diseases | interventions — Defibrillators, Implantable; Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRT=ON (Experimental): Cardiac Resynchronization Therapy activated.
  Interventions: Device: Implantable Cardioverter Defibrillator with Cardiac Resynchronization Therapy (BIOTRONIK Lumax HF-T CRT-D)
- CRT=OFF (Active Comparator): Cardiac Resynchronization Therapy deactivated.
  Interventions: Device: Implantable Cardioverter Defibrillator with Cardiac Resynchronization Therapy (BIOTRONIK Lumax HF-T CRT-D)

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator with Cardiac Resynchronization Therapy (BIOTRONIK Lumax HF-T CRT-D) — All patients will receive a commercially available BIOTRONIK Lumax HF-T CRT-D system with ICD back-up enabled. Patients will be randomized to CRT=ON or CRT=OFF.
  Other Names: Lumax HF-T CRT-D system

SUMMARY:
The EchoCRT trial evaluates the effects of Cardiac Resynchronization Therapy (CRT) on mortality and morbidity of subjects with heart failure due to left ventricular systolic dysfunction, already receiving optimized HF medication, with a narrow QRS width (< 130 ms) and echocardiographic evidence of ventricular dyssynchrony.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age or older.
* Understand the nature of the procedure.
* Give written informed consent.
* Willing and able to complete all testing required by the clinical protocol.
* Indication for an implantable cardioverter defibrillator (ICD).
* NYHA class III-IV within the last three months prior to enrollment and at baseline (at baseline only: also Stage C according to ACC/AHA guidelines).
* Stable optimal pharmacologic therapy for HF.
* An ejection fraction ≤ 35% within one year prior to enrollment and confirmed on the baseline echocardiogram.
* Increased left ventricular dimension, defined as LVEDD ≥ 55 mm.
* Resting QRS duration < 130 ms evidenced by a historical 12-lead ECG prior to enrollment and at baseline.
* Ventricular dyssynchrony assessed by echocardiography locally and confirmed by the echo core lab. One of the two following criteria has to be present to include the subject in the study:

  * Intra-left ventricular dyssynchrony measured by color Tissue Doppler Imaging (TDI) with an opposing wall delay of ≥ 80 ms in the 4-chamber or apical long-axis view.
  * Speckle-tracking radial strain septal-posterior wall delay ≥ 130 ms.

Exclusion Criteria:

* Implanted pacemaker or defibrillator with >10% ventricular pacing, as demonstrated by device statistics averaged over at least the last three months prior to enrollment.
* Women who are pregnant, lactating, or planning to become pregnant during the course of the trial.
* Bradycardia pacing indication.
* Surgically correctable primary valvular heart disease, i.e. aortic stenosis, torn cordae, or flail segment.
* Coronary artery bypass graft surgery or percutaneous coronary intervention (balloon and/or stent angioplasty) within the past 3 months prior to enrollment.
* Enzyme-positive myocardial infarction within the past 3 months prior to enrollment.
* Angiographic evidence of coronary disease, candidates for coronary revascularization likely to undergo coronary artery bypass graft surgery or percutaneous coronary intervention in the next 3 months.
* Irreversible brain damage from preexisting cerebral disease.
* Reversible non-ischemic cardiomyopathy such as acute viral myocarditis.
* Permanent second or third degree heart block.
* Chagas disease.
* Persistent or paroxysmal atrial fibrillation within one month prior to enrollment.
* Expected to receive heart transplantation within six months.
* Current inotropic therapy.
* Acutely decompensated heart failure.
* Contrast dye allergy and unable or unwilling to undergo pretreatment with steroids and/or diphenhydramine.
* Life expectancy of less than six months.
* Presence of any disease, other than the subject's cardiac disease associated with a reduced likelihood of survival for the duration of the trial, (e.g. cancer).
* Significant renal insufficiency defined as a serum creatinine > 2.5 mg/dL (> 221 µmol/L) within the last four weeks prior to enrollment..
* Liver failure, defined as three times the upper limit of normal for aminotransferases.
* Participation in any other clinical trial.
* Unable to return for follow-up visits due to distance from the clinic.
* Do not anticipate being a resident of the area for the scheduled duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1680 (Actual)
Dates: Start 2008-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Ruschitzka, MD, Study Chair — University of Zurich, Switzerland; Johannes Holzmeister, MD, Study Chair — University of Zurich, Switzerland; William Abraham, MD, Principal Investigator — Principal Investigator (USA) at The Ohio State University, OH, USA; Jagmeet Singh, MD, Principal Investigator — Principal Investigator (USA) at Massachusetts General Hospital, MA, USA
Locations (119):
- United States (59):
  - John Muir Medical Center, Concord, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Desert Cardiology, Rancho Mirage, California
  - University of California San Francisco, San Francisco, California
  - Cardiology Associates Medical Group, Ventura, California
  - Hartford Hospital, Hartford, Connecticut
  - Osceola Regional Medical Center, Kissimmee, Florida
  - University of Miami, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Tampa General Medical Center, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Saint Joseph's Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - St. Francis Medical Group, Indianapolis, Indiana
  - Community Heart and Vascular, Indianapolis, Indiana
  - Central Baptist Hospital, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Bay Regional Medical Center, Bay City, Michigan
  - Thoracic & Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Michigan Heart, P.C./ St. Joseph Mercy Hospital, Ypsilanti, Michigan
  - United Heart and Vascular Center, Saint Paul, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Kansas City Heart Foundation, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - St. Lukes-Roosevelt Hospital Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Sanger Heart & Vascular Institute, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Lindner Clinical Trial Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Richard M. Ross Heart Hospital, Columbus, Ohio
  - Promedica Northwest Ohio Cardiology Consultants, Toledo, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Lehigh Valley Heart Specialists, Allentown, Pennsylvania
  - Drexel Cardiology, Philadelphia, Pennsylvania
  - Jefferson Heart Institute, Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - South Carolina Heart Center, Columbia, South Carolina
  - The Stern Cardiovascular Center, Memphis, Tennessee
  - Cardiology Center of Amarillo, Amarillo, Texas
  - Texas Cardiac Arrhythmia, Austin, Texas
  - Cardiology Associates of Corpus Christi, Corpus Christi, Texas
  - University of Virginia, Charlottesville, Virginia
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Bon Secours Heart & Vascular Institute, Mechanicsville, Virginia
  - Virginia Cardiovascular Specialists, Richmond, Virginia
  - Bon Secours Heart & Vascular Institute, Richmond, Virginia
  - Cardiovascular Associates Ltd, Virginia Beach, Virginia
  - Kootenai Heart Clinics, Spokane, Washington
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin
- Australia (5):
  - Flinders Medical Center Adelaide, Adelaide
  - Princess Alexandra Hospital, Brisbane
  - St. Vincent's Hospital, Melbourne
  - Sir Charles Gairdner Hospital, Nedland
  - Royal Perth Hospital, Perth
- LKH Universitatsklinikum Graz, Graz, Austria
- Belgium (2):
  - OLV Hospital (OLV Ziekenhuis) Aalst, Aalst
  - Universitair Ziekenhuis Brussel, Brussels
- Canada (2):
  - UHN Toronto General Hospital, Toronto, Ontario
  - Edmonton Cardiology, Edmonton
- Czechia (3):
  - Olomouc University Hospital, Olomouc
  - IKEM - Institute for Clinical and Experimental Medicine, Prague
  - Na Homolce Hospital, Prague
- Denmark (4):
  - Aalborg Sygehus, Aalborg
  - Skejby Sygehus Aarhus, Aarhus
  - Rigshospitalet, Copenhagen
  - Gentofte Hospital, Hellerup
- France (3):
  - Nouvelles Cliniques Nantes, Nantes
  - CHU Pontchaillou de Rennes, Rennes
  - CHU Charles Nicolle, Rouen
- Germany (14):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Charite Campus Virchow Klinikum, Berlin
  - Judisches Krankenhaus Berlin, Berlin
  - Evangelisch-Freikirchliches Krankenhaus und Herzzentrum Brandenburg in Bernau, Bernau
  - Alfried Krupp Krankenhaus, Essen
  - Elisabeth-Krankenhaus Essen, Essen
  - Westdeutsches Herzzentrum Essen, Essen
  - Asklepios Klinik St. Georg Hamburg, Hamburg
  - Universitares Herzzentrum Hamburg GmbH, Hamburg
  - Universitatsklinikum Jena, Jena
  - Herzzentrum Leipzig GmbH, Leipzig
  - Klinikum Lüdenscheid, Lüdenscheid
  - St. Marien Hospital Lunen, Lünen
  - University Hospital of Magdeburg, Magdeburg
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Hadassah Medical Organization, Jerusalem
  - Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (4):
  - A.O.U. Consorziale Policlinico di Bari, Bari
  - A.O. Spedali Civili di Brescia, Brescia
  - P.O. Santa Maria di Loreto Nuovo, Naples
  - A.O.U. Maggiore della Carita, Novara
- Netherlands (2):
  - VU MC Amsterdam, Amsterdam
  - Leiden University Medical Center, Leiden
- Poland (2):
  - Instytut Kardiologii, Warsaw
  - 4 Wojskowy Szpital Kliniczny, Wroclaw
- Portugal (2):
  - Hospital Santa Maria de Lisboa, Lisbon
  - Hospital Santa Marta, Lisbon
- Spain (2):
  - University of Alicante General Hospital, Alicante
  - Hospital Clinic of Barcelona, Barcelona
- Switzerland (4):
  - Hopitaux Universitaires de Geneve, Geneva
  - CHU Vaudois Lausanne, Lausanne
  - Triemli Hospital (Stadtspital Triemli), Zurich
  - University of Zurich Hospital, Zurich
- United Kingdom (5):
  - University Hospitals of Coventry and Warwickshire, Coventry
  - Glenfield Hospital, Leicester
  - St. George's Hospital, London
  - St. Thomas' Hospital, London
  - Russells Hall Hospital, West Midlands

REFERENCES:
- [Derived] Varma N, Sogaard P, Bax JJ, Abraham WT, Borer JS, Dickstein K, Singh JP, Gras D, Holzmeister J, Brugada J, Ruschitzka F. Interaction of Left Ventricular Size and Sex on Outcome of Cardiac Resynchronization Therapy Among Patients With a Narrow QRS Duration in the EchoCRT Trial. J Am Heart Assoc. 2018 May 27;7(11):e009592. doi: 10.1161/JAHA.118.009592. PMID 29807890
- [Derived] Tayal B, Gorcsan J 3rd, Bax JJ, Risum N, Olsen NT, Singh JP, Abraham WT, Borer JS, Dickstein K, Gras D, Krum H, Brugada J, Robertson M, Ford I, Holzmeister J, Ruschitzka F, Sogaard P. Cardiac Resynchronization Therapy in Patients With Heart Failure and Narrow QRS Complexes. J Am Coll Cardiol. 2018 Mar 27;71(12):1325-1333. doi: 10.1016/j.jacc.2018.01.042. PMID 29566816
- [Derived] Steffel J, Varma N, Robertson M, Singh JP, Bax JJ, Borer JS, Dickstein K, Ford I, Gorcsan J 3rd, Gras D, Krum H, Sogaard P, Holzmeister J, Brugada J, Abraham WT, Ruschitzka F. Effect of Gender on Outcomes After Cardiac Resynchronization Therapy in Patients With a Narrow QRS Complex: A Subgroup Analysis of the EchoCRT Trial. Circ Arrhythm Electrophysiol. 2016 Jun;9(6):e003924. doi: 10.1161/CIRCEP.115.003924. PMID 27282848
- [Derived] Ruschitzka F, Abraham WT, Singh JP, Bax JJ, Borer JS, Brugada J, Dickstein K, Ford I, Gorcsan J 3rd, Gras D, Krum H, Sogaard P, Holzmeister J; EchoCRT Study Group. Cardiac-resynchronization therapy in heart failure with a narrow QRS complex. N Engl J Med. 2013 Oct 10;369(15):1395-405. doi: 10.1056/NEJMoa1306687. Epub 2013 Sep 2. PMID 23998714

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, baseline eligibility criteria were assessed (e.g. ventricular dyssynchrony, NYHA, QRS width, etc.) to qualify for implant. 1680 subjects were enrolled. 825 subjects did not qualify for implant and were exited from the study. 855 subjects qualified for implant. 821 subjects were successfully implanted. 809 subjects were randomized.
Groups:
- CRT=ON: Cardiac Resynchronization Therapy activated.
  Subject implanted with BIOTRONIK Lumax HF-T CRT-D system with ICD back-up enabled and randomized to CRT=ON.
- CRT=OFF: Cardiac Resynchronization Therapy deactivated.
  Subject implanted with BIOTRONIK Lumax HF-T CRT-D system with ICD back-up enabled and randomized to CRT=OFF.
Period: Overall Study
Arm/Group | CRT=ON | CRT=OFF
Started | 404 | 405
Completed | 0 | 0
Not Completed | 404 | 405
Not completed — Withdrawn due to study closure | 337 | 338
Not completed — Withdrawn prior to study closure | 13 | 28
Not completed — Lost to Follow-up | 5 | 6
Not completed — Vital status follow-up only | 3 | 3
Not completed — Death | 46 | 30

BASELINE CHARACTERISTICS:
Population: Baseline characterisics were analzed for the randomized population.
Groups:
- Total: Total of all reporting groups
Arm/Group | CRT=ON | CRT=OFF | Total
Number analyzed (Participants) | 404 | 405 | 809
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (12.9) | 58.3 (12.6) | 58.0 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 114 | 224
  Male | 294 | 291 | 585
Region of Enrollment [Number; unit: participants]
  Portugal | 4 | 3 | 7
  United States | 196 | 198 | 394
  Spain | 18 | 18 | 36
  Austria | 6 | 8 | 14
  Israel | 18 | 16 | 34
  United Kingdom | 19 | 18 | 37
  Switzerland | 11 | 11 | 22
  Italy | 4 | 4 | 8
  France | 10 | 11 | 21
  Czech Republic | 12 | 11 | 23
  Canada | 13 | 14 | 27
  Poland | 0 | 2 | 2
  Belgium | 6 | 6 | 12
  Australia | 12 | 11 | 23
  Denmark | 24 | 23 | 47
  Germany | 41 | 41 | 82
  Netherlands | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Composite Primary Endpoint: Number of Subjects With First Hospitalization for Worsening Heart Failure or Death
Description: The primary efficacy endpoint will evaluate the effect of CRT=ON versus CRT=OFF in time to event of a combined endpoint of all-cause mortality or first hospitalization for worsening heart failure.
Time Frame: From date of randomization until date of death from any cause or date of first hospitalization for worsening heart failure, whichever came first, assessed up to date of study exit, with a mean treatment duration of 1.6 years
Population: This analysis was carried out according to the intention-to-treat principle. Follow-up was censored at study closure, date of death, LVAD, heart transplant, withdrawal from the study, or loss to follow-up, whichever came first. 4 deaths in CRT OFF group and 1 death in CRT ON group were after LVAD/transplant and are not included in this analysis.
Measure: Number; unit: participants
Arm/Group | CRT=ON | CRT=OFF
Number analyzed (Participants) | 404 | 405
participants | 116 | 102

2. Primary Outcome: Number of Subjects That Underwent Implant Attempt Without System- or Implant-Related Complications (Complication-Free)
Description: The primary safety endpoint will evaluate the complication-free rate of the Lumax HF-T CRT-D devices in the narrow QRS subject population.
Time Frame: 6 months
Population: The primary safety endpoint included all subjects undergoing an implant procedure.
Measure: Number; unit: participants
Arm/Group | Subjects That Underwent an Implant Attempt
Number analyzed (Participants) | 855
participants | 766

3. Secondary Outcome: Rate of Hospitalizations for Worsening Heart Failure (Hospitalizations Per Subject-year)
Description: Evaluate the effects of CRT=ON compared to CRT=OFF on the rate of hospitalization for worsening heart failure (WHF).
Time Frame: Study duration from randomization to study exit
Measure: Number; unit: Hospitalizations per subj-yr
Arm/Group | CRT=ON | CRT=OFF
Number analyzed (Participants) | 404 | 405
Hospitalizations per subj-yr | 0.36 | 0.28

4. Secondary Outcome: New York Heart Association (NYHA) Classification Change
Description: Evaluate the effects of CRT=ON compared to CRT=OFF in relation to the change in NYHA classification.
  NYHA classes:
  Class I - Subjects with cardiac disease, but without resulting limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation,dyspnea, or anginal pain.
  Class II - Subjects with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III - Subjects with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain.
  Class IV - Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: 6 months
Population: Subjects with Baseline & 6-month NYHA classification. 18 subjects (9 CRT ON, 9 CRT OFF) that were in the study at least 6 months and that did not have 6-month NYHA data, had the most recent post-randomization NYHA inputted using the Last Observation Carried Forward (LOCF) principle.
Measure: Count of Participants; unit: Participants
Arm/Group | CRT=ON | CRT=OFF
Number analyzed (Participants) | 347 | 338
Participants
  Improved at least 1 Class | 213 | 185
  No Change | 116 | 141
  Deteriorated at least 1 Class | 18 | 12

5. Secondary Outcome: Change in Quality of Life (QOL) Scores From Baseline to 6-Month Follow-up
Description: Quality of Life was evaluated using the Minnesota Living with Heart Failure (MLHF) Quality of Life (QOL) Questionnaire.The questionnaire consists of 21 questions to measure the subjects' perception of how their HF and its treatment affected their ability to live as they wanted during the last month. The questions describe different ways in which some people are affected (i.e. physical, socioeconomic, and psychological impairments). If a question does not apply to a subject or is not related to their HF, then they can answer with a 0. If it does apply to them, then they can rate (from 1 to 5) how much it has affected them. From the 21 questions, the lowest possible total score is 0, and the highest possible total score is 105. A lower score is desirable. Therefore, a negative change in QOL score from baseline to 6 months represents an improvement in quality of life, while a positive change in QOL score from baseline to 6 months represents a worsening in quality of life.
Time Frame: Changes between baseline and 6 months
Population: Subjects with Baseline & 6-month QOL scores. 25 subjects (15 CRT ON, 10 CRT OFF) that were in the study at least 6 months and that did not have 6-month QOL data, had 3-month data inputted using the LOCF principle.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CRT=ON | CRT=OFF
Number analyzed (Participants) | 333 | 330
units on a scale | -12.1 (21.9) | -13.5 (21.4)

6. Secondary Outcome: Composite Score of Death, Hospitalization for Worsening Heart Failure and Change in Quality of Life (QOL)
Description: Evaluate the effects of CRT=ON compared to CRT=OFF in relation to a composite endpoint of all-cause mortality, hospitalization for worsening heart failure and change in the MLHF Quality of Life Questionnaire.
  This composite endpoint used a weighted scoring scale based on the African-American Heart Failure Trial (A-HeFT) study Endpoint Score. (Taylor, AL, Ziesche, S, Yancy, C, et al. Combination of Isosorbide Dinitrate and Hydralazine in Blacks with Heart Failure. N Engl J Med 2004; 351:2049-57.)
  Composite Endpoint Scoring:
  Vital Status:
  Death (-3),
  Survival to end of trial (0),
  Hospitalization:
  1st hospitalization for HF (-1),
  No hospitalization (0),
  QOL score:*
  Improvement by ≥ 10 units (+2),
  Improvement by 5-9 units (+1),
  Change by < 5 units (0),
  Worsening by 5-9 units (-1),
  Worsening by ≥ 10 (-2).
  Possible total score -6 to +2.
  *QOL score details are provided in Secondary Outcome Measure 5.
Time Frame: Composite of death, worsening heart failure hospitalization (up to 24 months), and change in QOL (at 6 months)
Population: Subjects with a potential of 24 months of follow-up.
Measure: Mean (Standard Deviation); unit: Composite score
Arm/Group | CRT=ON | CRT=OFF
Number analyzed (Participants) | 163 | 163
Composite score | -1.6 (1.9) | -1.5 (1.6)

7. Secondary Outcome: Number of Subjects With All-cause Mortality
Description: Evaluate the all-cause mortality rate between the CRT=ON compared to CRT=OFF group.
Time Frame: From date of randomization up to date of study exit, with a mean treatment duration of 1.6 years
Measure: Count of Participants; unit: Participants
Arm/Group | CRT=ON | CRT=OFF
Number analyzed (Participants) | 404 | 405
Participants | 45 | 26

ADVERSE EVENTS:
Time Frame: Study duration from date of implant to date of study exit, with a mean implant duration of 1.7 years
Description: Subjects could have more than one event. Other adverse event data includes data from non-serious adverse events.
Arm/Group | CRT=ON | CRT=OFF
All-Cause Mortality (participants affected / at risk) | 45/404 | 26/405
Serious Adverse Events (participants affected / at risk) | 259/404 | 221/405
Other Adverse Events (participants affected / at risk) | 300/404 | 274/405
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT=ON (N=404) | CRT=OFF (N=405)
Worsening heart failure (Cardiac disorders) | 101 (213) | 93 (181)
Atrial arrhythmia (Cardiac disorders) | 27 (34) | 25 (35)
Ventricular arrhythmia (Cardiac disorders) | 26 (36) | 22 (29)
Chest pain (Cardiac disorders) | 16 (31) | 21 (26)
Other cardiovascular (Cardiac disorders) | 18 (21) | 17 (20)
Dyspnea (Cardiac disorders) | 16 (16) | 11 (12)
Coronary artery disease (Cardiac disorders) | 13 (13) | 10 (11)
Infection (Infections and infestations) | 58 (77) | 45 (54)
Gastrointestinal disorder (Gastrointestinal disorders) | 43 (68) | 28 (41)
Other noncardiovascular (General disorders) | 40 (54) | 36 (55)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 14 (27) | 22 (38)
Renal disorder (Renal and urinary disorders) | 28 (38) | 16 (19)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 25 (32) | 15 (18)
Nervous system disorder (Nervous system disorders) | 13 (16) | 5 (5)
ICD lead (Cardiac disorders) | 23 (26) | 13 (13)
Lead for right atrial pacing (Cardiac disorders) | 18 (21) | 5 (5)
Lead for left ventricular pacing (Cardiac disorders) | 18 (21) | 4 (4)
Implantation related (Surgical and medical procedures) | 17 (19) | 16 (18)
Hypotension (Cardiac disorders) | 11 (14) | 9 (9)
Angina (Cardiac disorders) | 7 (8) | 12 (13)
Peripheral vascular disease (Cardiac disorders) | 6 (8) | 10 (12)
Syncope (Cardiac disorders) | 8 (8) | 7 (9)
Cardiac arrest (Cardiac disorders) | 11 (13) | 3 (3)
Myocardial infarction (Cardiac disorders) | 6 (6) | 6 (8)
Anemia (Cardiac disorders) | 5 (9) | 4 (4)
Stroke (Cardiac disorders) | 6 (7) | 6 (6)
Pulmonary embolism (Cardiac disorders) | 5 (5) | 5 (7)
Transischemic attack (Cardiac disorders) | 6 (6) | 4 (4)
Thrombosis (Cardiac disorders) | 3 (3) | 5 (6)
Fluid accumulation (Cardiac disorders) | 5 (7) | 1 (1)
Pulmonary edema (Cardiac disorders) | 5 (5) | 2 (3)
Cardiac catheterization (Cardiac disorders) | 5 (5) | 2 (2)
Cardiovascular medication related (Cardiac disorders) | 3 (3) | 4 (4)
Dizziness (Cardiac disorders) | 4 (4) | 3 (3)
Pleural effusion (Cardiac disorders) | 4 (4) | 2 (2)
Valvular heart disease (Cardiac disorders) | 4 (5) | 1 (1)
Abdominal Aortic Aneurysm (Cardiac disorders) | 3 (3) | 2 (2)
Edema (Cardiac disorders) | 1 (1) | 3 (3)
Increased INR (Cardiac disorders) | 2 (3) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Dilated cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Ischemic cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Weight gain (Cardiac disorders) | 2 (2) | 0 (0)
Fatigue (Cardiac disorders) | 1 (1) | 0 (0)
Endocrine (Endocrine disorders) | 12 (13) | 4 (6)
Cancer (General disorders) | 5 (5) | 10 (13)
Traumatic injury (General disorders) | 11 (12) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 3 (4)
Hepatic (Hepatobiliary disorders) | 1 (2) | 2 (2)
Fatigue (General disorders) | 3 (3) | 0 (0)
Device related (Cardiac disorders) | 6 (6) | 9 (10)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT=ON (N=404) | CRT=OFF (N=405)
Worsening heart failure (Cardiac disorders) | 29 (32) | 29 (34)
Atrial arrhythmia (Cardiac disorders) | 39 (44) | 35 (43)
Ventricular arrhythmia (Cardiac disorders) | 33 (39) | 25 (29)
Chest pain (Cardiac disorders) | 20 (21) | 29 (32)
Dyspnea (Cardiac disorders) | 20 (27) | 30 (32)
Hypotension (Cardiac disorders) | 27 (28) | 27 (30)
Dizziness (Cardiac disorders) | 21 (25) | 14 (15)
Edema (Cardiac disorders) | 21 (23) | 15 (16)
Non-cardiovascular (General disorders) | 203 (602) | 201 (548)
Implant Procedure (Surgical and medical procedures) | 31 (33) | 41 (46)
ICD lead (Cardiac disorders) | 28 (34) | 6 (6)
Lead for left ventricular pacing (Cardiac disorders) | 49 (55) | 10 (11)

LIMITATIONS AND CAVEATS:
Endpoint results should be interpreted with caution and take into consideration the early study closure and subsequent reduction in sample size (809 vs. 1258) and events (218 vs. 381). These changes impact the statistical power of the findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No